CLINICAL TRIAL: NCT02441478
Title: Co-operative Behavior and Decision-making in Frontal Lobe Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL14-0269
Record Dates: First submitted 2015-04-03; First posted 2015-05-12 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Frontal Lobe Epilepsies
Keywords: cooperative behavior, therapy adherence, fMRI
MeSH Terms: conditions — Epilepsy, Frontal Lobe; Cooperative Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental)
  Interventions: Radiation: functional magnetic resonance imaging exam
- Controls (Active Comparator)
  Interventions: Radiation: functional magnetic resonance imaging exam

INTERVENTIONS:
Radiation: functional magnetic resonance imaging exam
  Other Names: fMRI exam

SUMMARY:
Epilepsy is a frequent neurological disorder with about a third of patients having seizures despite treatment. At least some of these seizures can be linked to a low compliance and therapy adherence of patients. Compliance is defined as "the extent to which a person's behavior (in terms of taking medication, following diets, or executing life style changes) coincides with medical or health advice". Therapy adherence of patients suffering from epilepsy is low with reported rates between 30 and 50%, although adherence to anticonvulsive drug therapy is critical for effective disease management and low therapy adherence is associated to higher mortality in epilepsy. The reasons for low therapy adherence are still a matter of research. Some known factors influencing compliance in epilepsy are related to its chronic nature, but others seem to lie in a complex interaction between psychiatric comorbidity and an impairment of neural systems underlying behavior. Furthermore, therapy adherence rests a variable difficult to measure, especially in epileptic patients where classical tools such as questionnaires and electronic monitoring devices have been shown to be imprecise. It has been argued that the term 'compliance' should be replaced by 'co-operative behavior' and non-compliance can therefore be interpreted as troubled co-operative behavior. This behavioral approach offers the potential of using tools and methods of the latest developments in behavioral neuroscience. Neuroeconomics, a scientific field on the border of psychology, economics and neuroscience, has used economic game paradigms in order to operationalize cooperative behavior and to identify several brain areas by functional brain imaging that have been linked to social co-operative behavior. The majority of these brain areas are located in the frontal cortex [ventromedial frontal/orbitofrontal cortex, and rostral anterior cingulate cortex. Epilepsies originating in the frontal lobe are subsumed under the term "frontal lobe epilepsy" (FLE) and represent 20-30% of all partial seizures and 25% of all refractory focal epilepsies referred to epilepsy surgery.

The investigator's project plans to study compliance and cooperative behavior of patients suffering from frontal lobe epilepsies through a neuroeconomic approach by (1) comparing the behavior of these patients in the prisoners' dilemma game to the behavior of age-, gender-, and education-matched healthy controls, (2) correlation of game behavior to brain activation measured by functional magnetic resonance imaging in both patients and healthy controls and (3) studying the link between cooperative behavior to compliance captured by pill counts and questionnaires.

ELIGIBILITY:
Inclusion Criteria (Patients):

* Age between 18 and 50
* Diagnosis of frontal lobe epilepsy
* Written consent to participate
* Right-handed
* Hospital Anxiety and Depression Scale Score under 10
* Obsessive Compulsive Inventory Score under 40
* Sufficient language skills
* Social insurance

Inclusion criteria (controls):

* Age between 18 and 50
* Written consent to participate
* Right-handed
* Hospital Anxiety and Depression Scale Score under 10
* Obsessive Compulsive Inventory Score under 40
* Sufficient language skills
* Social insurance

Exclusion Criteria (Patients):

* Seizures types other than epileptic (psychogenic etc.)
* Mental retardation
* Epilepsies other than FLE
* Other known neurological diseases
* Hospital Anxiety and Depression Scale Score over 10
* Obsessive Compulsive Inventory Score over 40
* Pregnancy
* non-MRI suitable transplants (cardiac pacemaker etc.), claustrophobia, orthopedic diseases that prevent lying in the scanner
* During exclusion period of other studies
* No social insurance

Exclusion criteria (controls)

* History of neurological or psychiatric diseases
* Hospital Anxiety and Depression Scale Score over 10
* Obsessive Compulsive Inventory Score over 40
* Medication other than contraceptives
* Pregnancy
* non-MRI suitable transplants (cardiac pacemaker etc.), claustrophobia, orthopedic diseases that prevent lying in the scanner
* Major perceptive impairments
* During exclusion period of other studies
* No social insurance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Social cooperative behavior as measured by the prisoners' dilemma game | 1 day
  The prisoners' dilemma game (PDG; Trivers, 1971) is a well-studied game derived from economic game theory that has been used extensively to quantify and study cooperative behavior. The two players in the game can choose between two moves, either "co-operate" or "defect". If both players co-operate, they both receive the reward R. If one player defects, while the other one co-operates, then the defector receives the payoff T while the co-operative player receives the payoff S. If both players defect, they both receive the payoff P. (T > R > P > S).

SECONDARY OUTCOMES:
Blood-oxygen-level dependent signal during the Prisoners' dilemma game | 1 day
  Whole brain analysis of correlation between behavior in the PDG (prisoners' dilemma game) and brain activation as measured by the BOLD (blood-oxygen-level dependent) signal captured through functional MRI as well as group differences between patients and controls.
Neuropsychological profile | 1 day
  analysis of neuropsychological testing of (working) memory, attention, theory-of-mind and executive functions.
Pill counts | 1 day
  Pills taken and not-taken during the study period will be counted as a variable of therapy adherence.
Scores acquired by questionnaire | 1 day
  Several questionnaires to cover beliefs about therapy adherence will be applied.
Scores acquired by questionnaire | 1 day
  questionnaire to cover beliefs about medicines will be applied
Scores acquired by questionnaire | 1 day
  questionnaire to cover beliefs about trust towards physicians and medications will be applied

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Background] Javor A, Ciumas C, Ibarrola D, Ryvlin P, Rheims S. Social cognition, behaviour and therapy adherence in frontal lobe epilepsy: a study combining neuroeconomic and neuropsychological methods. R Soc Open Sci. 2019 Aug 28;6(8):180850. doi: 10.1098/rsos.180850. eCollection 2019 Aug. PMID 31598216